CLINICAL TRIAL: NCT00276276
Title: An Open-Label, Multicentre, Randomised, Phase III Comparator Study of Active Symptom Control Alone or in Combination With Oral Topotecan in Patients With Relapsed Resistant SCLC
Brief Title: Active Symptom Control Alone Or In Combination With Oral Topotecan In Patients With Relapsed Resistant Small Cell Lung Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 104864/478
Record Dates: First submitted 2006-01-11; First posted 2006-01-13 (Estimated); Last update posted 2013-04-15 (Estimated); Status verified 2012-11

CONDITIONS: Lung Cancer, Small Cell
Keywords: relapsed; lung cancer; resistant; small cel; topotecan (HYCAMTIN)
MeSH Terms: conditions — Small Cell Lung Carcinoma; Recurrence; Lung Neoplasms | interventions — Topotecan

INTERVENTIONS:
Drug: topotecan

SUMMARY:
The purpose of this study is to find out if giving oral HYCAMTIN to patients with relapsed small cell lung cancer benefits them. The study will compare how long patients live when they are given therapy to make them feel better (active symptom control) to the length of time patients live when they are also receiving oral HYCAMTIN.

ELIGIBILITY:
Inclusion Criteria:

* Received one prior chemotherapy regimen only.
* Documented partial or complete response to first-line therapy.
* Documented relapse of limited or extensive SCLC at least 45 days after the cessation of first-line chemotherapy.
* Not considered suitable for further intravenous chemotherapy.
* Considered to have adequate bone marrow reserve.
* Performance Status of 0, 1 or 2.

Exclusion Criteria:

* Pregnant or lactating.
* Received more than one prior regimen of chemotherapy.
* Uncontrolled vomiting.
* Brain metastases.
* Active uncontrolled infection.
* Received previous treatment with HYCAMTIN.
* Received an investigational product within 30 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 141
Dates: Start 2000-11

PRIMARY OUTCOMES:
Overall survival

SECONDARY OUTCOMES:
Time to response, response rate, time to disease progression

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (15):
- Bulgaria (3):
  - GSK Investigational Site, Pleven
  - GSK Investigational Site, Plovdiv
  - GSK Investigational Site, Varna
- Hungary (5):
  - GSK Investigational Site, Budapest
  - GSK Investigational Site, Csorna
  - GSK Investigational Site, Hungary
  - GSK Investigational Site, Miskolc
  - GSK Investigational Site, Törökbálint
- GSK Investigational Site, Breda, Netherlands
- GSK Investigational Site, Moscow, Russia
- Ukraine (2):
  - GSK Investigational Site, Donetsk
  - GSK Investigational Site, Lviv
- United Kingdom (3):
  - GSK Investigational Site, Chelmsford, Essex
  - GSK Investigational Site, Glasgow, Lanarkshire
  - GSK Investigational Site, Sutton, Surrey

REFERENCES:
- [Background] O'Brien ME, Ciuleanu TE, Tsekov H, Shparyk Y, Cucevia B, Juhasz G, Thatcher N, Ross GA, Dane GC, Crofts T. Phase III trial comparing supportive care alone with supportive care with oral topotecan in patients with relapsed small-cell lung cancer. J Clin Oncol. 2006 Dec 1;24(34):5441-7. doi: 10.1200/JCO.2006.06.5821. PMID 17135646